CLINICAL TRIAL: NCT07069023
Title: The Effect of Breath Exercise and Reiki Application on Tiredness and Nausea and Vomiting Management in Oncology Patients; Randomised Controlled Study
Brief Title: Tiredness and Nausea and Vomiting Management in Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BCU1259; Reıkı and Oncology Patients (Registry Identifier: Reıkı and Oncology Patients)
Record Dates: First submitted 2025-05-21; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Fatigue; Nausea
Keywords: Breath exercise; reiki application; tiredness; nausea; vomiting
MeSH Terms: conditions — Neoplasms; Fatigue; Nausea; Vomiting | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study employed a three-group experimental design involving a breathing exercise group, a Reiki group, and a control group. Participants in the intervention groups received sessions twice a week for six weeks, while the control group received no intervention. Data were collected at three points: pre-test (week 1), mid-test (week 3), and post-test (week 6), using validated instruments. These assessments aimed to measure changes over time and compare group differences. Ethical approval was obtained, and informed consent was secured from all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reiki group (Active Comparator): Oncology patients with nausea, vomiting and fatigue received reiki throughout the treatment.
  Interventions: Other: breathing exercise group; Other: reiki group
- breathing exercise group (Active Comparator): Oncology patients with nausea, vomiting and fatigue were given breathing exercises throughout the treatment.
  Interventions: Other: breathing exercise group; Other: reiki group

INTERVENTIONS:
Other: breathing exercise group — Oncology patients with nausea, vomiting and fatigue were given breathing exercises throughout the treatment.
  Other Names: control group
Other: reiki group — Oncology patients with nausea, vomiting and fatigue received reiki throughout the treatment.

SUMMARY:
This randomised controlled trial will investigate the effects of breathing exercises and Reiki on fatigue and nausea-vomiting symptoms in oncology patients. Data will be collected through face-to-face interviews using structured forms before the start of chemotherapy. To account for possible losses, 20 patients will be included in each intervention group.

DETAILED DESCRIPTION:
Objective: This study aims to investigate the effects of breathing exercises and reiki on symptoms of fatigue, nausea, and vomiting.

Experimental procedure: This randomised controlled trial will be conducted to investigate the effects of breathing exercises and reiki on symptoms of fatigue, nausea, and vomiting in oncology patients. Data will be collected using data collection forms during approximately 30-minute face-to-face interviews immediately before patients begin chemotherapy treatment. Considering that there may be case losses during the study, it was decided to include 20 patients in each group.

ELIGIBILITY:
Inclusion Criteria: Patients who volunteered to participate in the study, were diagnosed with cancer, had symptoms of nausea-vomiting and fatigue, were literate, could communicate, did not have a diagnosis of mental or psychiatric illness, were not hearing or visually impaired, were 18 years of age or older, and were not receiving antiemetic treatment.

-

Exclusion Criteria:Patients with any other disease related to the gastrointestinal system, any other disease or condition that would prevent them from performing the exercises to be performed for the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Individual Introductory Information Form | 6 WEEKS
  It was consists of questions such as socio-demographic characteristics such as age, marital status, chronic diseases, disease history, and type, stage, metastasis status, metastasis site, treatment status, nausea and vomiting
Hirai Cancer Fatigue Scale | 6 WEEKS
  The scale measures fatigue in cancer patients and is 5-point Likert type. The minimum value of the scale is 15 and the maximum value is 75. High scores on the scale indicate increased fatigue and low scores indicate decreased fatigue.The Cronbach Alpha value of the original scale was found to be 0.943.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Temiz, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol